CLINICAL TRIAL: NCT05342974
Title: A Pilot Study of Atorvastatin as a Potential Adjunct to Misoprostol for Termination of Pregnancy
Brief Title: Atorvastatin as a Potential Adjunct to Misoprostol for Termination of Pregnancy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00148011
Record Dates: First submitted 2022-03-22; First posted 2022-04-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Abortion Early
Keywords: abortion; medical abortion; atorvastatin; misoprostol
MeSH Terms: interventions — Atorvastatin; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Atorvastatin followed by misoprostol (Experimental): Oral dose of atorvastatin (80 mg) to be taken daily for seven days followed by misoprostol (800 mcg) on day 8. A second dose of misoprostol will occur 24 hours after the first dose if no significant bleeding (more than a regular period) has occurred.
  Interventions: Drug: Atorvastatin; Drug: Misoprostol

INTERVENTIONS:
Drug: Atorvastatin — Oral dose of atorvastatin (80 mg) to swallow at the clinic in the presence of a study provider with additional 6 doses (80 mg each) of atorvastatin to administer at home once daily for the next six days. These 6 pills should be taken orally. Return to the clinic for a follow-up visit approximately 3, 8 and 10 days after enrollment visit. At these visits, trained study clinician will evaluate abortion status using ultrasound and blood draw. At 8-day visit post-enrollment, 800 mcg of misoprostol will be provided to be taken vaginally or allowed to dissolve between cheek and tongue for 30 minutes, within 24 hours of the visit. At the final clinic visit, 10 days post-enrollment, if the termination of pregnancy has failed, standard abortion care at the clinic will be offered. A final phone call to assess any side effects, need for medical care or complications will occur 30 days after enrollment.
Drug: Misoprostol — On Study Day 8, participant will be provided will two doses of misoprostol 800 mcg for vaginal or buccal use. Participant will take a single dose of misoprostol on study day 8 (± 1 day), and be instructed to take an additional 800 mcg vaginal or buccal misoprostol if no significant bleeding consistent with passage of tissue (heavier than a menses) has occurred within 24 hours of first misoprostol dose.

SUMMARY:
Medication abortion is a way of ending a pregnancy using pills. The current FDA-approved regimen for medication abortion uses mifepristone and misoprostol. This study is testing whether a different medication, atorvastatin, followed by misoprostol, can be used to end a pregnancy. Participants at 35-49 days of pregnancy will receive an oral dose of atorvastatin (80 mg) to swallow at the clinic as well as taking atorvastatin (80 mg) daily for six additional days, with a return to clinic on day 8 after initial visit to take a dose of misoprostol (800 mcg). Additionally, follow-up visits will occur on approximately days 3, 8 and 11 for a clinician to perform an ultrasound to see if the abortion is complete.

DETAILED DESCRIPTION:
Safe and legal abortion is an important part of reproductive health. Medication abortion using a combination of mifepristone and misoprostol is recognized worldwide as the gold standard for early medication abortion. Finding another medication that replace mifepristone would benefit both those who need abortions and providers around the world. Atorvastatin might be one drug that could do this. It is a statin that is commercially available in many countries.

Goal: To evaluate the safety and effectiveness of a user-friendly atorvastatin-misoprostol regimen

Primary Objective: Successful interference in pregnancy progress, decreases in measurable human chorionic gonadotrophin (HCG) hormone, or an end of pregnancy (prior to misoprostol use) within seven days of starting atorvastatin (80 mg per day for seven days).

Sample Size: 30 patients

Location: Recruitment of all participants and data collection will take place at Planned Parenthood Association of Utah.

Study Population: People presenting to the study site for medical abortion who have an intrauterine pregnancy visible on ultrasound with a single fetus ≤ 49 days gestational age.

Study Procedures:

STUDY DAY 1 (at clinic) The pregnancy will be confirmed to be 35- 49 days gestational age through transvaginal ultrasound. Baseline data will be collected including pregnancy symptoms and prior medical pregnancy history. Atorvastatin will be started at 80 mg per day for 7 days (first dose taken in clinic). The remaining six doses will be provided to take at home. A blood draw will occur to measure HCG hormone levels.

STUDY DAY 3 (at clinic) Participants will come to clinic, and blood will be drawn to measure HCG hormone levels and a transvaginal ultrasound will occur to monitor pregnancy status.

STUDY DAY 8 (at clinic, day after final day of atorvastatin) A transvaginal ultrasound will be completed to view pregnancy status. Participant will be provided two doses of misoprostol (800 mcg) that can be taken buccally (inserted into cheeks until they dissolve - approximately 30 minutes) or inserted vaginally. The second dose will be taken at home if participant does not experience bleeding that indicates end of pregnancy (heavier than a standard period) within 24 hours.

STUDY DAY 9-11 FOLLOW-UP (at clinic):

In clinic, an exam will be conducted to confirm that the abortion has been completed and to review symptoms that have occurred. If the abortion is not complete, a standard abortion with uterine evacuation will be provided within the week to complete the abortion.

EXTENDED FOLLOW-UP (by text, email, or phone):

30 days after starting the study, participants will be contacted to document any side effects or any needed medical care related to the abortion or complications from the abortion. This will occur through phone or email. These follow up data will address any lasting side effects, need for additional medical care, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* A pregnancy confirmed as 35-49 days gestational age through transvaginal ultrasound
* Seeking termination of pregnancy
* Speak English or Spanish
* Willing to potentially delay abortion for 1-2 weeks
* Willing and able to comply with study protocol and accept that the study regimen may not successfully terminate the pregnancy thus a uterine aspiration would be required to complete the abortion.
* Willing to delay contraception until completion of abortion

Exclusion Criteria:

* People with pregnancy over 49 days gestational age
* Twin or higher multiple pregnancy
* Medical contraindications to medical abortion per the mifepristone U.S. Food and Drug Administration label
* Confirmed or suspected ectopic pregnancy
* Vaginal bleeding in current pregnancy
* Pregnancy of unknown location
* IUD or contraceptive implant in place
* History of allergy to atorvastatin or misoprostol
* History of myositis
* Currently taking or planning on taking medications during the study that interact with HMG co-A reductase inhibitors (e.g., diltiazem, erythromycin, azoles, gemfibrozil or another fibrate)
* Unable to return for clinic-based follow-up
* Currently breastfeeding
* Already taking an HMG co-A reductase inhibitor [37] or plan to take one outside the study drug during the trial (Fluvastatin, lovastatin, pitavastatin, pravastatin, simvastatin, fluvastatin, lovastatin, pitavastatin, pravastatin, rosuvastatin, simvastatin or rosuvastatin.
* Unable to swallow pills

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Interference in pregnancy progress | Within 7 days of initiating atorvastatin (80 mg per day)
  This is a dichotomous outcome that includes interference in pregnancy progress by any of the following: ultrasound markers as measured by transvaginal ultrasonographic loss of embryonic cardiac activity or abnormal ultrasonographic growth over seven day period, decreases in human chorionic gonadotrophin measures through insufficient rise in quantitative HCG will be considered any of the following: a decrease or increase of less than 50% in quantitative HCG from day 1 to 3; a decrease or increase of less than 100% in quantitative HCG from day 3 to 7, or expulsion of pregnancy prior to misoprostol use.

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, MPH, Principal Investigator — University of Utah
Locations (1):
- Planned Parenthood Association of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD may be shared with other researchers with a legitimate and proven interest in conducting further analyses.
Time Frame: 5 years from completion of study
Access Criteria: Requests made to the PI via email will be considered.